CLINICAL TRIAL: NCT04155060
Title: The Prognostic Value of Lactate is Different Among Septic Patients With or Without Diabetes Mellitus
Brief Title: The Prognostic Value of Lactate is Different Among Septic Patients
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROMPT
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Sepsis; Diabetes Mellitus
Keywords: hyperlactatemia
MeSH Terms: conditions — Sepsis; Diabetes Mellitus; Hyperlactatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DM group , non-DM group: Septic patients were divided into the DM group and non-DM group, based on their comorbidity
- high lactate group,low lactate group: high lactate group (lactate > 2 mmol/L) and low lactate group (lactate ≤ 2 mmol/L), according to the admission lactate level.

SUMMARY:
Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection. Early diagnosis of sepsis and identification of more severe sepsis is important to improve the outcomes .Therefore, reliable markers are required to early identify the high-risk patients. Currently, lactate is widely applied as the marker for evaluating the severity of sepsis and for outcome predicting. DM affects lactate balance and raised baseline lactate. The objective of this study was to compare the different prognostic value of admission lactate for sepsis patients with or without DM.

DETAILED DESCRIPTION:
Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection. Early diagnosis of sepsis and identification of more severe sepsis is important to improve the outcomes .Therefore, reliable markers are required to early identify the high-risk patients.

Currently, lactate is widely applied as the marker for evaluating the severity of sepsis and for outcome predicting.Nevertheless, the value of lactate for predicting sepsis is still controversial.The reasons for the different cutoff value may be due to the fact that sepsis is a heterogeneous disease which has already been defined by a number of clinical, laboratory and radiologic criteria, rather than specific pathologic findings. Therefore, we hypothesized that the discrepancy clinical value of lactate may be resulted from the heterogeneous feature of sepsis.

DM affects lactate balance and raised baseline lactate. The objective of this study was to compare the different prognostic value of admission lactate for sepsis patients with or without DM.

ELIGIBILITY:
Inclusion Criteria:18 years or older, informed consent signed, admission serum lactate level obtained, and admission to the hospital with sepsis or septic shock diagnosis.

-

Exclusion Criteria:congenital metabolic and psychiatric diseases and clinical data deficiency.

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic patients were recruited with lactate level obtained, and admission to the intensive care unit (ICU) .
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome was 28-day mortality | up to at least 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No